CLINICAL TRIAL: NCT04495699
Title: Treatment of Asymptomatic Renal Calculi in Recurrent UTIs: a Prospective Observational Cohort Study
Brief Title: Asymptomatic Renal Calculi in Recurrent Urinary Tract Infections
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of British Columbia (Other); University of California, San Diego (Other); Mayo Clinic (Other); Massachusetts General Hospital (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Ryan Hsi, Associate Professor, Department of Urology, Vanderbilt University Medical Center
Other Study IDs: 0000000
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Urinary Tract Infections; Kidney Stone
Keywords: Urinary Tract Infection; Kidney Stones; Urolithiasis
MeSH Terms: conditions — Urinary Tract Infections; Kidney Calculi; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observation: Patients who elect to have observation of their asymptomatic stones as part of usual care will be followed. Note that there is no randomization, the decision to treat or not treat a stone is made in the usual clinical fashion by the patient in consultation with their surgeon.
- Stone treated: Patients who elect to have intervention of their asymptomatic stones as part of usual care will be followed. Note that there is no randomization, the decision to treat or not treat a stone is made in the usual clinical fashion by the patient in consultation with their surgeon.
  Interventions: Other: None - observational

INTERVENTIONS:
Other: None - observational — If the patient elects to have their stone treated, it will be treated in the usual most clinically appropriate fashion (Shockwave lithotripsy, ureteroscopy, or percutaneous nephrolithotomy). All types of treatment will be analyzed together.
  Groups: Stone treated

SUMMARY:
This study will assess patients who have recurrent urinary tract infections and kidney stones which are not blocking the kidney or causing other problems. Currently, we don't know if taking out these stones will improve recurrent urinary tract infections or not. Patients will make a decision with their surgeon about removing or monitoring their stone(s). Whether or not their infections continue with surgery or monitoring will be noted, and this information may help to inform future treatment decisions. The purpose of this study is to assess if treatment of these asymptomatic stones affects the rate of recurrent urinary tract infections.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are common and have a large burden of disease at the population level. This study will assess the effectiveness of removing kidney stones in patients who have recurrent UTIs.

The role of upper urinary tract calculi in UTIs is not well understood. Although there is some evidence that some metabolic stones, such as calcium oxalate, can harbor bacteria, it is not known if this is clinically significant or if these contribute to clinical infections.

This study aims to advance the level of evidence in the treatment of non-obstructing urolithiasis in the context of recurrent UTIs.

The aim of this study is to:

1. Assess the effects of treatment of non-obstructing upper urinary tract calculi on recurrent UTIs in the first prospective observational trial in this area

Patients who meet inclusion criteria will make a decision about treating their asymptomatic stones or not with their surgeon as per usual clinical care. The primary outcome will be the rate of recurrent urinary tract infections for patients, comparing patients who did and did not have their stones treated.

Patient data is securely stored in de-identified fashion in REDCAP database, following all the secure protocols of the institutions involved. The recruitment goal is 80 patients based on power calculations to detect the effect size. Statistical analysis will be performed between the two groups, with t-test used for normally distributed numerical data and fisher's exact or chi-square tests for categorical data.

ELIGIBILITY:
Inclusion Criteria (all of the following):

* recurrent UTIs, defined as 3 positive urine cultures of specific organisms with symptoms within 12 months (or 2 positive cultures with symptoms within 6 months) prior to clinical assessment
* non-obstructing renal stone(s) on imaging within 6 months of initial visit

Exclusion Criteria:

* age < 18 years
* pregnancy
* hydronephrosis or evidence of obstruction
* presence of a foreign body in urinary tract (e.g. Foley, ureteral stent, nephrostomy tube) at the time of UTI diagnosis
* concurrent bladder calculi
* Urinary diversion or previous surgery involving segments of bowel interposed into the urinary tract (ileal conduit, ileal ureter etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent UTIs and asymptomatic renal calculi.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Recurrent urinary tract infections | 12 months
  • Number of UTIs, defined as positive urine culture (>10^5 CFU/mL of a specific organism) with symptoms. If having had surgical intervention for the stones, we will count a UTI during >30days and <1year after intervention so that it is not attributed to the intervention

SECONDARY OUTCOMES:
Time to first UTI | up to 12 months
  Time from first visit to first UTI, defined as above
Pyelonephritis/urosepsis | up to 12 months
  Incidence of pyelonephritis/urosepsis
Incidence of complications from intervention within 30 days | 30 days
  Clavien-Dindo complications, ER visits, readmissions, infections within 30 days, non-elective repeat interventions (eg for obstructing fragments)
Incidence of further intervention for stones | 12 months
  any further stone interventions required
Stone analysis correlation with rUTI | 12 months
  Correlation between primary outcome and stone analysis
Stone free vs not stone free correlation with rUTI | 12 months
  Correlation between stone free status after intervention and recurrent UTI
Correlation of selected demographic factors with rUTI | 12 months
  Correlation between baseline demographic parameters and recurrent UTIs (including include age, sex, bacteria type, previous sequelae from UTIs, previous sequelae from stones, comorbidities including diabetes mellitus, obesity, hypertension, and immunosuppression, creatinine, total stone burden, location of stones, stone composition, stone culture, post-intervention stone free rate, and 24-h urine parameters if available)
Number free from recurrent UTIs | 12 months
  Number patients free of recurrent UTIs at 1 year, defined as 3 positive urine cultures (>105 CFU/mL of a specific organism) with symptoms in 1 year, or 2 in 6 months. If having had surgical intervention for the stones, we will count a UTI during >30days and <1year after intervention so that it is not attributed to the intervention
Number free from any UTI | 12 months
  Number of patients free from any UTI at one year, as defined above
Crossover from observation to intervention | 12 months
  Patients on observation and decide to seek treatment after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hsi, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (5):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Vancouver General Hospital/University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anger J, Lee U, Ackerman AL, Chou R, Chughtai B, Clemens JQ, Hickling D, Kapoor A, Kenton KS, Kaufman MR, Rondanina MA, Stapleton A, Stothers L, Chai TC. Recurrent Uncomplicated Urinary Tract Infections in Women: AUA/CUA/SUFU Guideline. J Urol. 2019 Aug;202(2):282-289. doi: 10.1097/JU.0000000000000296. Epub 2019 Jul 8. PMID 31042112
- [Background] Agarwal DK, Krambeck AE, Sharma V, Maldonado FJ, Westerman ME, Knoedler JJ, Rivera ME. Treatment of non-obstructive, non-struvite urolithiasis is effective in treatment of recurrent urinary tract infections. World J Urol. 2020 Aug;38(8):2029-2033. doi: 10.1007/s00345-019-02977-3. Epub 2019 Oct 23. PMID 31646382
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Barr-Beare E, Saxena V, Hilt EE, Thomas-White K, Schober M, Li B, Becknell B, Hains DS, Wolfe AJ, Schwaderer AL. The Interaction between Enterobacteriaceae and Calcium Oxalate Deposits. PLoS One. 2015 Oct 8;10(10):e0139575. doi: 10.1371/journal.pone.0139575. eCollection 2015. PMID 26448465
- [Background] Cai T, Mazzoli S, Mondaini N, Meacci F, Nesi G, D'Elia C, Malossini G, Boddi V, Bartoletti R. The role of asymptomatic bacteriuria in young women with recurrent urinary tract infections: to treat or not to treat? Clin Infect Dis. 2012 Sep;55(6):771-7. doi: 10.1093/cid/cis534. Epub 2012 Jun 7. PMID 22677710
- [Background] Flannigan RK, Battison A, De S, Humphreys MR, Bader M, Lellig E, Monga M, Chew BH, Lange D. Evaluating factors that dictate struvite stone composition: A multi-institutional clinical experience from the EDGE Research Consortium. Can Urol Assoc J. 2018 Apr;12(4):131-136. doi: 10.5489/cuaj.4804. Epub 2017 Dec 22. PMID 29319486
- [Background] Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Dis Mon. 2003 Feb;49(2):53-70. doi: 10.1067/mda.2003.7. PMID 12601337
- [Background] Geerlings SE. Clinical Presentations and Epidemiology of Urinary Tract Infections. Microbiol Spectr. 2016 Oct;4(5). doi: 10.1128/microbiolspec.UTI-0002-2012. PMID 27780014
- [Background] Griebling TL. Urologic diseases in america project: trends in resource use for urinary tract infections in men. J Urol. 2005 Apr;173(4):1288-94. doi: 10.1097/01.ju.0000155595.98120.8e. PMID 15758784
- [Background] Omar M, Abdulwahab-Ahmed A, Chaparala H, Monga M. Does Stone Removal Help Patients with Recurrent Urinary Tract Infections? J Urol. 2015 Oct;194(4):997-1001. doi: 10.1016/j.juro.2015.04.096. Epub 2015 Apr 30. PMID 25936865